CLINICAL TRIAL: NCT05215301
Title: Assessment of Multidimensional Voice Program (MDVP) Parameters in Occupational and Non-occupational Voice Users: a Secondary Data Analysis
Brief Title: Assessment of Multidimensional Voice Program (MDVP) Parameters in Workers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Other Study IDs: THT003
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Voice Disorders; Occupational Problems; Work-related Illness
Keywords: Multidimensional Voice Disorder; Voice Quality; Occupational Voice Users
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Occupational Voice Users: Workers who uses voice extensively during work falls under occupational voice users (e.g. singers, actors, radio announcer, teacher, translator, lawyer). The grouping were made based on references from The Union of the European Phoniatricians
  Interventions: Diagnostic Test: Multidimensional Voice Program
- Non-occupational Voice Users: Those who didn't use voice extensively during work falls under non-occupational voice users (motorcycle drivers, daily labor, administrative workers)
  Interventions: Diagnostic Test: Multidimensional Voice Program

INTERVENTIONS:
Diagnostic Test: Multidimensional Voice Program — MDVP (Multidimensional Voice Program) is a computerized acoustic analysis used to analyze sound quality using various parameters. Multidimensional Voice Program (MDVP) 4500 produced by Kay Elemetric Corp was used for voice evaluation.
  Research subjects were asked to make a vowel sound /"a"/ using the same tone and intensity as the subject's daily speech. The researcher will give an example before letting the research subject tries. Voice recording was done using a microphone connected to a computer with the MDVP program. Voice recording was done in a quiet room for at least 3 seconds with a microphone distance of 10 cm from the mouth of the research subject. The recorded sound will be directly analyzed with the MDVP program. Sound recording was done 3 - 5 times, and the best sound acoustic analysis results were used for the study.
  Other Names: Acoustic Phonation Program; Kay Elemetric Corp MDVP 4500

SUMMARY:
MDVP (Multidimensional Voice Program) has several parameters that can assess voice quality objectively, including Base Frequency (F0), Jitter, Shimmer, NHR (Noise to Harmonic Ratio), VTI (Voice Turbulence Index), and ATRI (Amplitude Tremor Intensity Index). MDVP may provide an objective yet non-invasive and comfortable alternative to assess voice quality - and to some extent, diagnose voice-related abnormalities. The utilization of MDVP in clinical settings is quite common but using it concerning occupational health is rare, especially in Indonesia. No study had reported usage of MDVP to assess voice quality in any occupational voice user group or reported a thorough comparison of MDVP parameters between occupational and non-occupational voice users. With an increase in the realization that voice can be an essential occupational modality, MDVP may become a practical alternative modality in assessing voice quality and occupational-related voice injury in clinical settings. This study will determine any association between occupational voice users and their MDVP parameters from medical records and the MDVP database in Dr Cipto Mangunkusumo Hospital, Jakarta. The study also tries to see whether there is any value in using MDVP to assess voice quality in workers.

DETAILED DESCRIPTION:
Data will be extracted from the MDVP database and hospital medical records. The MDVP database consists of patients examined with MDVP in the Department of ORL-HNS' Larynx-Pharynx clinic of Dr. Cipto Mangunkusumo Hospital, Jakarta.

Voice evaluation for all patients in Dr. Cipto Mangunkusuomo Hospital was done using the Multidimensional Voice Program (MDVP) 4500 produced by Kay Elemetrics Corp installed on a personal computer. The patients were asked to emit vocal sounds /" a "/ using the tone and intensity of everyday speech. The physicians are obliged to give an example first. The patient's voice was then recorded using a microphone connected to a computer with the MDVP program. Sounds were recorded in a quiet room for at least 3 seconds with the microphone 10 cm from the patient's mouth. The MDVP program will directly analyze the recorded sound. Sound recording is done 3 - 5 times, and the best sound acoustic analysis results are used as the final result. The results are then kept in the program's database inside the computer.

Patients who attend the Larynx-Pharynx clinic for MDVP evaluations are usually those who comes for post-treatment monitoring (e.g., post-laryngoplasty), had been diagnosed with a voice disorders, and or by personal or physicians' request. There are various reasons why patients are being assigned to MDVP evaluations - and all of this information will be gathered and used as a consideration during data analysis. For the sake of practicality, the researcher will only extract MDVP data from the past five years. Other considerations will be made to ensure that the data extracted will represent a reliable comparison between occupation status and how it affects MDVP parameters (see more in "Criteria for subjects"). The study will use total sampling, where all available data that fits the inclusion criteria will be used for analysis.

Inclusion criteria

* Patients had their medical records and MDVP data available in dr. Cipto Mangunkusumo Hospital, Jakarta
* Patients are active workers in Indonesia on the time of MDVP evaluation
* Patients are above the age of 18
* Patients can be either an occupational or non-occupational voice users Exclusion criteria
* Patients with incomplete occupational data
* Patient with incomplete MDVP results

Data obtained from the database will be evaluated in SPSS v20 software and analysed to produce descriptive and inferential statistics. The inferential statistics will consist of univariate analysis and bivariate analysis (between two variables). All numeric data will be tested for normal distribution using Kolmogorov-Smirnov.

Univariate analysis will be done to see the average, distribution, and frequency of all variables/outcomes which include the participants' demographic information and MDVP parameters. MDVP parameters will be presented as mean score with its standard deviation (or median with range). Bivariate analysis will be done to evaluate the significance between occupational or non-occupational users to their MDVP parameters. Differences between groups will be assessed using independent samples t-test (parametric) or Mann-Whitney (non-parametric). If possible, multivariate analysis will also be conducted using Chi-Square or Fischer test depending on the data distributions.

ELIGIBILITY:
Inclusion Criteria:

* Patients had their medical records and MDVP data available in dr. Cipto Mangunkusumo Hospital, Jakarta
* Patients are active workers in Indonesia on the time of MDVP evaluation
* Patients are above the age of 18
* Patients can be either an occupational or non-occupational voice users

Exclusion Criteria:

* Patients with incomplete occupational data
* Patient with incomplete MDVP results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be extracted from the MDVP database and hospital medical records. The MDVP database consists of patients examined with MDVP in the Department of ORL-HNS' Larynx-Pharynx clinic of Dr. Cipto Mangunkusumo Hospital, Jakarta.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
F0 (Fundamental Frequency) | 3 minutes minimal
  Average fundamental frequency for the vocalization measured in Hz
Jitter | 3 minutes minimal
  Jitter refers to a disruption in sound wave frequencies caused by a lack of control over the vibrations of the vocal cords.
Shimmer | 3 minutes minimal
  Shimmer percent gives an evaluation in percent of the variability of the peak-to-peak amplitude within the analyzed voice samples. It represents the relative period-to-period (very short-term) variability of the peak-to-peak amplitude
NHR (Noise to Harmonic Ratio) | 3 minutes minimal
  Noise-to-harmonic ratio is an average ratio of energy of the in-harmonic components in the range 1500-4500 Hz to the harmonic components energy in the rage 70-4500 Hz. It is a general evaluation of the noise present in the vocalization
ATRI (Amplitude Tremor Intensity Index) | 3 minutes minimal
  Amplitude tremor intensity index shows (in percent) the ratio of the amplitude of the most intensive low-frequency amplitude-modulating component (amplitude tremor) to the total amplitude of the analyzed voice signal.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhael Yosia, MD, Principal Investigator — Department of Community Medicine, Faculty of Medicine Universitas Indonesia; Dewi S Soemarko, MD, Study Chair — Department of Community Medicine, Faculty of Medicine Universitas Indonesia; Marsen Isbayuputra, MD, Study Chair — Department of Community Medicine, Faculty of Medicine Universitas Indonesia; Syahrial M Hutauruk, MD, Study Chair — Department of ORL-HNS, Faculty of Medicine Universitas Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will be kept in Cipto Mangunkusumo General Hospital and will only be shared upon official request to the hospital.

REFERENCES:
- [Result] Kosztyla-Hojna B, Rogowski M, Ruczaj J, Pepinski W, Lobaczuk-Sitnik A. An analysis of occupational dysphonia diagnosed in the North-East of Poland. Int J Occup Med Environ Health. 2004;17(2):273-8. PMID 15387083
- [Result] Feder RJ. Varix of the vocal cord in the professional voice user. Otolaryngol Head Neck Surg. 1983 Aug;91(4):435-6. doi: 10.1177/019459988309100417. PMID 6415594
- [Result] Godino-Llorente JI, Osma-Ruiz V, Saenz-Lechon N, Cobeta-Marco I, Gonzalez-Herranz R, Ramirez-Calvo C. Acoustic analysis of voice using WPCVox: a comparative study with Multi Dimensional Voice Program. Eur Arch Otorhinolaryngol. 2008 Apr;265(4):465-76. doi: 10.1007/s00405-007-0467-x. Epub 2007 Oct 9. PMID 17922287